CLINICAL TRIAL: NCT04146688
Title: Nonverbal Communication in Aged People With and Without Neurodegenerative Disease: Study of Sensorimotor Synchronization to Music
Brief Title: Nonverbal Communication in Aged People
Acronym: MAMUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: France Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_35; 2017-A03543-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-09; First posted 2019-10-31 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Alzheimer Disease
Keywords: Music; Communication; Emotion; Behavior; Neurodegeneration disease
MeSH Terms: conditions — Alzheimer Disease; Communication; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with neurodegenerative disease (Active Comparator): Patients with neurodegenerative disease (AD or related disease)
  Interventions: Other: Music Balance Board
- People with no neuropathological disease (Active Comparator)
  Interventions: Other: Music Balance Board

INTERVENTIONS:
Other: Music Balance Board — The SSM is measured with an innovative tool (Music Balance Board) developed at the University of Ghent (Belgium) and specially designed to record the movements of the elderly in a natural and comfortable position This chair is equipped with a tablet and sensors that record the movements of the hand and body during the SSM to a musical sequence. The analysis will focus on the difference between the participant's striking and the beat of the music measured using this chair.

SUMMARY:
Musical interventions improve the emotional state of patients with Alzheimer's disease (AD) while having a positive impact on the caregiver's well-being. However, the factors that could be responsible for this positive effect remain unknown. Among these, the sensory-motor synchronization (SMS) of movements to the musical rhythm, frequently observed during musical activities and possible up to the advanced stages of AD, could modulate the emotional state. Several recent studies have shown that rhythmic training (or SMS) influences the organism at the motor, cognitive and social levels while activating the cerebral reward circuit. This action that generates pleasure also facilitates non-verbal emotional expression. However, the conditions that modulate SMS and their relationship to nonverbal communication, emotional, behavioral and cognitive state have not yet been studied in healthy or pathological elderly.

ELIGIBILITY:
Inclusion Criteria:

Cases : Patients with neurodegenerative disease (AD or related disease)

* Native French Language
* Corrected auditory and/or visual deficiency
* Right-handed
* Image rights consent signed by the patient Controls: People with no neuropathological disease
* Native French Language
* Corrected auditory and/or visual deficiency
* Right-handed
* Image rights consent signed by the control

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
measure of consistency (oppositive of variability) | Baseline, before SMS task
  measure of consistency (oppositive of variability) of the response corresponding to the length of a vector going from 0 (bad) to 1(very good response).
  This measure is completed by another measure of asynchrony.
measure of asynchrony. | Baseline, before SMS task
  The asynchrony assess the accuracy of the movements in ms. If the participant anticipated the tap relative to the musical beat, the value is negative, if the participant delayed the tap, the value is positive. A perfect tap is 0 in this case

SECONDARY OUTCOMES:
Measurement of the Music Balance Board (cf. primary outcome) during music in the presence of a real experimenter | Baseline, before SMS task
  measure the quantity of movements derived from the variation of weight on the sensors below the platform in millivolts (mV)
Measurement of the Music Balance Board (cf. primary outcome) during music in the presence of a virtual experimenter; | after SMS task, an average after 45 min
  measure the quantity of movements derived from the variation of weight on the sensors below the platform in millivolts (mV)
Measurement of the Music Balance Board (cf. primary outcome) during metronome in the presence of a real experimenter | after SMS task, an average after 45 min
  measure the quantity of movements derived from the variation of weight on the sensors below the platform in millivolts (mV)
Measurement of the Music Balance Board (cf. primary outcome) during metronome in the presence of a virtual experimenter. | after SMS task, an average after 45 min
  measure the quantity of movements derived from the variation of weight on the sensors below the platform in millivolts (mV)
Decoding of non-verbal behaviors during the synchronization task | after SMS task, an average after 45 min
  Decoding of non-verbal behavior during the synchronization task (rhythmic movements of the head, lips and lower limbs, visual contact) in duration (duration of the behavior/duration of the Condition expressed in seconds) by blind evaluators in the membership group.
Intensity of body movements (quantity of motion) | after SMS task, an average after 45 min
  Intensity of body movements (quantity of motion) recorded by the motion sensors connected to the chair on which the patient sits.
  recorded during the SSM test and a filmed interview
STAI Anxiety Scale Score | through study completion, an average of 2 hours
  The State-Trait Anxiety Inventory (STAI) is a self-questionnaire, developed by Spielberger (7) and validated in French. It has 20 questions, assessing the subject's usual emotional state. A score is calculated, ranging from 20 to 80, a high score indicating the presence of anxiety.
Decoding of the frequency (number of behaviors / duration of the condition) of the facial expressions | through study completion, an average of 2 hours
  the facial expressions based on videoscopic recordings of the synchronization task and a short interview (5min) by blind evaluators of the home group.
Scale of Assessment of Daily Activities | through study completion, an average of 2 hours
  The ADLs used measure of functional ability is the Katz Activities of Daily Living Scale (Katz et al., 1963; Katx, 1983). In this scale, the set of tasks assessed are bathing, dressing, transferring, using the toilet, continence, and eating.
Scale of Instrumental Activities of Daily Living | through study completion, an average of 2 hours
  The Lawton IADL Scale takes approximately 10 to 15 minutes to administer. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning)
Neuropsychiatric Inventory (NPI) subscales Impact on the workload of the caregiver. | through study completion, an average of 2 hours
  total NPI score is defined as the sum of the individual category scores. Higher scores on NPI indicate a more frequent and/or severe presence of neuropsychiatric behavioral changes. The following domains will be included in the subscore: Depression/Dysphoria, Anxiety, Apathy/Indifference, Irritability/Lability, Agitation/Aggression, and Disinhibition.
mini-mental state examination (MMSE) score | through study completion, an average of 2 hours
  The Mini-Mental State Examination (MMSE) is a brief 30-point questionnaire test that is used to screen for cognitive impairment.
  Scores on a scale range from 0 - 30. Scores 23 and below are indicative of problems.
Concentration of cortisol from saliva samples | Once, at Day 1, baseline
  measure the saliva cortisol before and after the synchronization task

CONTACTS AND LOCATIONS:
Overall Officials: François Puissieux, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital les Bateliers, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No